CLINICAL TRIAL: NCT05428527
Title: Real-world Clinical Benefit Evaluation in Breast Cancer Patients With Pharmaceutical Interventions for Cancer-related Fatigue
Status: Completed | Type: Observational
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Taichung Veterans General Hospital (Other); E-Da Cancer Hospital (Unknown); Chang Gung Memorial Hospital, Taipei (Unknown); Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other); China Medical University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital, Keelung (Unknown)
Responsible Party: Principal Investigator, Ming-Shen Dai, Chief of Department of Oncology, National Defense Medical Center, Taiwan
Other Study IDs: CRF-NHI01
Record Dates: First submitted 2022-06-13; First posted 2022-06-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cancer-related Fatigue
Keywords: Cancer-related Fatigue; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients with Cancer-related fatigue treatment: Breast cancer patients who approved to use NHI to pay for Cancer-related fatigue treatment drug

SUMMARY:
This retrospective study is to collect and analyze the data from medical records within the period that breast cancer patient is receiving NHI-covered CRF treatment. This study will evaluate the clinical use, fatigue improvement, and treatment satisfaction of breast cancer patients with CRF treatment.

DETAILED DESCRIPTION:
This is a single arm, multicenter, and retrospective study. About 200 breast cancer patients' data from medical records are expected to collect and analyze in this retrospective study. The data collection from medical records of breast cancer patients who approved to use NHI to pay for CRF treatment drug will include the demographic information, disease characteristics and cancer treatment information, fatigue score by visual analog fatigue scale, fatigue clinical global impression, CRF pharmacological treatment record, hematological lab data, ECOG, cancer drug compliance record, overall clinical evaluation after CRF treatment by physicians and patient's expectation to continue CRF treatment etc. Data of three return visits (i.e. at the time of before CRF treatment, after 4 times of CRF treatment and CRF treatment completed) per patient will be collected from medical records to analysis within the period that patient is receiving NHI-covered CRF treatment.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients who approved to use NHI to pay for cancer-related fatigue treatment drug

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: breast cancer patients who approved to use NHI to pay for cancer-related fatigue treatment drug
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue Improvement | through study completion, an average of 4 months

SECONDARY OUTCOMES:
The Level of Fatigue Clinical Global Impression-Improvement | through study completion, an average of 4 months
Physician Satisfaction Degree of Overall Clinical Evaluation | 1 time, average of 4 months after baseline (at the end of study)
Patient Expectation Rating of Continuous Cancer-Related Fatigue Treatment | 1 time, average of 4 months after baseline (at the end of study)
ECOG Change | through study completion, an average of 4 months
Weight Change | through study completion, an average of 4 months
Hematological Lab Data Change | through study completion, an average of 4 months
The Incidence of Cancer Treatent Delay | through study completion, an average of 4 months
The Incidence of Cancer Treatent Dose Modification | through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Locations (9):
- Taiwan (9):
  - E-Da Cancer Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided